CLINICAL TRIAL: NCT00909168
Title: Induction, Consolidation and Intensification Therapy for Patients Younger Than 66 Years With Previously Untreated CD33 Positive Acute Myeloid Leukemia (AML)
Acronym: MYFLAI07
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Udine, Italy (Other)
Responsible Party: Principal Investigator, CANDONI ANNA, Division of Hematology, SM MISERICORDIA HOSPITAL, University Hospital, Udine, Italy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYFLAI07
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Induction chemotherapy; Fludarabine; Gemtuzumab Ozogamicin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Cytarabine; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Efficacy of FLAIMy (Experimental)
  Interventions: Drug: FLAIMy - Fluda, Ida, Ara-C, Mylotarg

INTERVENTIONS:
Drug: FLAIMy - Fluda, Ida, Ara-C, Mylotarg — FLUDARABINE: 25 mg/m2/day, 250 FS in 30', start h 9 - 1, 2, 3, 4, 5
  ARABINOSYL-CYTOSINE (Cytarabine): 2 g/m2/day, 500 FS in 3 h, start h 13 - 1, 2, 3, 4, 5
  IDARUBICIN: 10 mg/m2/day, 100 FS in 1 h, start h 16 - 1, 3, 5
  GEMTUZUMAB OZOGAMICIN (Mylotarg): 5 mg, single dose 500 FS in 4 h - 6

SUMMARY:
This is a prospective, open, non-randomized, non-controlled, phase II, clinical trial for treatment of newly diagnosed AML patients, younger than 66 years.

Trial is based on:

* INDUCTION: FLAI + Gemtuzumab-Ozogamicin (FLAI-GO).
* CONSOLIDATION: Intermediate dose AraC + IDA (IDAC+IDA) +/- one course of high dose AraC (HDAC)
* INTENSIFICATION: Allo-BMT, ASCT
* MAINTENANCE: AraC

  a) Primary endpoints:
* Feasibility, Efficacy (CR+PR rate) and Toxicity of FLAI + Gemtuzumab-Ozogamicin.
* RFS, DFS and OS.

  b) Secondary endpoints:
* Evaluation of Minimal Residual Disease by WT1 (and other biologic markers) expression and monitoring.
* Evaluation of prognostic clinical relevance of biological features at onset.
* Feasibility and outcome of consolidation with BMT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* WHO PS grade 0-2 (Appendix B) or Karnofsky > 70.
* AML according to the new WHO criteria, i.e., % of BM blasts ≥ 20%. NB. this % should be assessed on a BM aspiration or on a BM biopsy
* All FAB subtypes except M3.
* CD33 positivity (> 20%). It is mandatory to perform an immunotyping of the BM blasts in particular the determination of CD33 positivity, which will be used as a inclusion factor.
* Previously untreated (except ≤ 14 days of Hydroxyurea) primary or secondary AML (including AML after MDS).
* Adequate renal and liver function, i.e., creatinine < 2 mg/dl and bilirubin, ALT/AST ≤ 3 times the upper limit of normal.
* Written informed consent

Exclusion Criteria:

* Blast crisis of chronic myeloid leukemia.
* AML supervening after other myeloproliferative diseases.
* AML de novo or secondary previously pretreated.
* Concomitant malignant disease.
* Active central nervous system (CNS) leukemia.
* Active uncontrolled infection [NB severe systemic infection should be excluded].
* Concomitant severe cardiovascular disease, i.e., arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease.
* Cardiac ejection fraction of 50% or less.
* Severe pulmonary dysfunction (CTC grade 3-4).
* Severe concomitant neurological or psychiatric disease.
* History of alcohol abuse.
* HIV positivity.
* Pregnancy.
* Man and woman not agreeing to the adequate contraceptive precautions during study period and for at last 24 months after stop of therapy.
* Any psychological, familiar, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Feasibility, Efficacy (CR+PR rate) and Toxicity of FLAI + Gemtuzumab-Ozogamicin. | one year
RFS, DFS and OS. | one year

SECONDARY OUTCOMES:
Evaluation of Minimal Residual Disease by WT1 (and other biologic markers) expression and monitoring. | one year
Evaluation of prognostic clinical relevance of biological features at onset. | one year
Feasibility and outcome of consolidation with BMT. | one year

CONTACTS AND LOCATIONS:
Overall Officials: ANNA CANDONI, MD, Study Director — UUNIVERSITY HOSPITAL, UDINE, ITALY
Locations (1):
- University Hospital, Udine, Udine, Italy, Italy

REFERENCES:
- [Derived] Candoni A, Papayannidis C, Martinelli G, Simeone E, Gottardi M, Iacobucci I, Gherlinzoni F, Visani G, Baccarani M, Fanin R. Flai (fludarabine, cytarabine, idarubicin) plus low-dose Gemtuzumab Ozogamicin as induction therapy in CD33-positive AML: Final results and long term outcome of a phase II multicenter clinical trial. Am J Hematol. 2018 May;93(5):655-663. doi: 10.1002/ajh.25057. Epub 2018 Mar 2. PMID 29396857